CLINICAL TRIAL: NCT00170716
Title: Safety and Effectiveness of Targeted Sub-Threshold Epidural Cortical Stimulation Delivered Concurrent With Rehabilitation Activities to Enhance Motor Recovery in Patients Suffering From Upper Extremity Hemiparesis Following a Stroke
Brief Title: Safety and Effectiveness of Cortical Stimulation in the Treatment of Stroke Patients With Upper Extremity Hemiparesis
Acronym: EVEREST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northstar Neuroscience (Industry)
Responsible Party: VP Clinical Affairs, Northstar Neuroscience
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V0267
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Stroke; Hemiparesis
Keywords: Motor Cortex Electrical Stimulation; Ischemic Stroke; Upper Extremity Hemiparesis; Rehabilitation; Motor Recovery; Functional MRI
MeSH Terms: conditions — Stroke; Paresis; Ischemic Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator)
  Interventions: Other: Rehabilitation
- Investigational (Experimental)
  Interventions: Device: Cortical Stimulation and rehabilitation

INTERVENTIONS:
Device: Cortical Stimulation and rehabilitation — Cortical stimulation is provided concomitantly with rehabilitation therapy. Rehabilitation is for 2.5 hrs per day for 26 days over a period of 6 weeks.
  Other Names: Renova-ST Cortical Stimulation System
  Arms: Investigational
Other: Rehabilitation — Rehabilitation is for 2.5 hrs per day for 26 days over a period of 6 weeks.
  Other Names: Post-stroke rehabilitation.
  Arms: Control

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of cortical stimulation delivered concurrent with rehabilitation activities to enhance motor recovery in patients suffering from hemiparesis affecting the upper extremity following a stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of serious, long-term disability in the United States. According to the American Stroke Association, the prevalence of stroke in the U.S. is approximately 4.8 million with approximately 700,000 additional strokes occurring annually. The 2001 overall death rate for stroke was 58%. Of those who survive, 30 to 50 percent do not regain functional independence, 15 to 30 percent are permanently disabled, and 20% require institutional care at three months after onset.

The most common neurological deficit among these stroke survivors, and thus a substantial contributor to post-stroke disability, is a motor weakness on one (hemiparesis) side of the body. Presently, the only treatment available for patients with motor deficits is rehabilitative therapy. However, many patients are not responsive to standard rehabilitative therapy or achieve a less than satisfactory improvement in function.

The primary objective of this study is to determine the safety and effectiveness of targeted sub-threshold epidural cortical stimulation delivered concurrent with rehabilitation activities to enhance motor recovery in patients suffering from hemiparesis (a motor weakness in one half of the body) affecting the upper extremity (shoulder, arm, wrist, hand) following a stroke. In addition to evaluating changes from baseline level, safety and efficacy measures will be compared to patients who undergo the same rehabilitation activities but without cortical stimulation. The two study groups will be compared to determine the degree to which motor function of the affected limb can be improved beyond rehabilitation alone by epidural stimulation of a targeted cortical region.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have an ischemic stroke.
* Moderate to moderately severe upper-extremity hemiparesis.
* Aged 21 years or older.

Exclusion Criteria:

* Primary hemorrhagic stroke.
* Any additional stroke associated with incomplete motor recovery.
* Any neurologic or physical condition impairing function of the target extremity.
* History of seizure disorder.
* History of spinal cord injury, traumatic brain injury, or spontaneous subdural or epidural hematoma that has resulted in a neurologic deficit.
* Contraindication to magnetic resonance (MR) imaging.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2004-09; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Arm Motor Fugl-Meyer (AMFM) score | Follow Up Week 4
Arm Motor Ability Test (AMAT) score | Follow Up Week 4

SECONDARY OUTCOMES:
Box and Block Test score | Follow Up Week 4
Stroke Specific Quality of Life (SSQOL) score | Follow Up Week 4
Serious adverse event rate | Follow up week 4 and 6 months

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Colorado Neurological Institute & Swedish Medical Center, Englewood, Colorado
  - University of Florida, Jacksonville, Jacksonville, Florida
  - Emory Clinic, Atlanta, Georgia
  - Northwestern University Medical Center and the Rehabilitation Institute of Chicago, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Spaulding Rehabilitation Center and Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - State University of New York Upstate Medical Center, Syracuse, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Health Sciences Center at Houston, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Swedish Health Services, Seattle, Washington

REFERENCES:
- [Background] Brown JA, Lutsep H, Cramer SC, Weinand M. Motor cortex stimulation for enhancement of recovery after stroke: case report. Neurol Res. 2003 Dec;25(8):815-8. doi: 10.1179/016164103771953907. PMID 14669524
- [Background] Cramer SC, Benson RR, Himes DM, Burra VC, Janowsky JS, Weinand ME, Brown JA, Lutsep HL. Use of functional MRI to guide decisions in a clinical stroke trial. Stroke. 2005 May;36(5):e50-2. doi: 10.1161/01.STR.0000163109.67851.a0. Epub 2005 Apr 14. PMID 15831835
- [Background] Brown JA, Lutsep HL, Weinand M, Cramer SC. Motor cortex stimulation for the enhancement of recovery from stroke: a prospective, multicenter safety study. Neurosurgery. 2006 Mar;58(3):464-73. doi: 10.1227/01.NEU.0000197100.63931.04. PMID 16528186
- [Derived] Levy RM, Harvey RL, Kissela BM, Winstein CJ, Lutsep HL, Parrish TB, Cramer SC, Venkatesan L. Epidural Electrical Stimulation for Stroke Rehabilitation: Results of the Prospective, Multicenter, Randomized, Single-Blinded Everest Trial. Neurorehabil Neural Repair. 2016 Feb;30(2):107-19. doi: 10.1177/1545968315575613. Epub 2015 Mar 6. PMID 25748452
- See also: Related Info — http://www.northstarneuro.com/clinicaltrials/patient_motorrecovery.asp
- See also: Related Info — http://www.northstarneuro.com/clinicaltrials/physician_motorrecovery.asp